CLINICAL TRIAL: NCT01052220
Title: Improving Blood Pressure Control in End-Stage Renal Disease Through a Supportive-Educative Nursing Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Zorica Kauric-Klein, Assistant Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0904007039; HIC# 2009-94 (Other: William Beaumont Hospital, Royal Oak Michigan); 020-2009 (Other: Davita Clinical Research)
Record Dates: First submitted 2010-01-19; First posted 2010-01-20 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Hypertension; Hemodialysis
Keywords: Hypertension; Blood Pressure; End Stage Renal Disease; Hemodialysis; Interdialytic Weight Gain; Self-Regulation
MeSH Terms: conditions — Hypertension; Kidney Failure, Chronic; Self-Control | interventions — Organizational Objectives; Reinforcement Machine Learning; Professional Autonomy

STUDY DESIGN:
Intervention Model Description: Participants were randomized to intervention group of standard care.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BP Education and Self Regulation of BP (Experimental): The intervention will consist of 3 phases: 1) BP education sessions, 2) 12 week intervention and 3) 30 day post intervention follow-up period. The participants in the treatment group will received a BP educational session at baseline and were asked to monitor and record home BP daily, 24 hour fluid intake and complete a salt intake check-lists twice weekly for 12 weeks.
  The PI made weekly visits with the intervention participants in the HD unit to review BP and fluid logs and salt check lists with the participant to determine if predetermined goals for BP control were attained. When goals related to BP control are met, positive verbal reinforcement will be given to the participant. When goals related to BP control are not met, further exploration and problem solving will be done.
  Interventions: Behavioral: BP education and BP self-regulation; Behavioral: Supportive Educative Nursing Intervention
- Usual Care (No Intervention): Participants in the usual care group did not receive the intervention but continued to receive their standard care in the hemodialysis unit which involved follow-up by the medical provider and BP medication adjustments as needed. .

INTERVENTIONS:
Behavioral: BP education and BP self-regulation — The intervention will consist of 3 phases: 1) BP education sessions, 2) 12 week intervention and 3) 30 day post intervention follow-up period. The participants in the treatment group will be asked to monitor and record home BP daily, 24 hour fluid intake and complete a salt intake check-lists twice weekly for 12 weeks.
  The PI will visit weekly with the intervention participants in the HD unit. to review BP and fluid logs and salt check lists with the participant to determine if predetermined goals for BP control were attained. When goals related to BP control are met, positive verbal reinforcement will be given to the participant. When goals related to BP control are not met, further exploration and problem solving will be done.
  Other Names: Home Blood Pressure Monitoring; Goal Setting; Reinforcement
  Arms: BP Education and Self Regulation of BP
Behavioral: Supportive Educative Nursing Intervention — BP Education, BP, salt and fluid monitoring, BP goal-setting, and reinforcement
  Other Names: Self-regulation
  Arms: BP Education and Self Regulation of BP

SUMMARY:
The major purpose of this quantitative study is to determine if a 3 month supportive educative nursing intervention incorporating Blood Pressure (BP) education and BP, salt and fluid monitoring, in addition to goal setting and reinforcement will improve BP control in a chronic end-stage renal disease population.

DETAILED DESCRIPTION:
120 Participants will be recruited for the study. The participants will be randomized to either an intervention or control group. Randomization will occur according to the Hemodialysis (HD)unit the participant dialyzes at. The intervention will consist of 3 phases: 1) education sessions, 2) 12 week intervention and 3) 30 day post intervention follow-up period. The intervention group will receive two 15 minute individual education sessions conducted by the research coordinator in the HD unit.

The objectives of session 1 are: 1) to explain the underlying pathophysiology and associated risks of high BP in HD, 2) to identify the goals that can improve BP control and 3) to describe the role of self-regulation in changing behavior related to BP control. The objectives of Session 2 include: to provide and demonstrate correct participant use of home BP monitors, correct recording of home BPs, 24 hr fluid recall and salt intake checklists. The participants will also receive educational pamphlets on methods to improve salt and fluid restrictions.

The participants in the treatment group will be asked to monitor and record their home BP, salt and fluid intake weekly for 12 weeks. The research coordinator will have weekly 10 to 15 minute visits with the intervention participants in the HD unit. The PI will review BP and fluid logs and salt check lists with the participant to determine if predetermined goals for BP control were attained. When goals related to BP control are met, positive verbal reinforcement will be given to the participant. When goals related to BP control are not met, further exploration and problem solving will be done.

The control group will receive standard care which involves BP monitoring and medication adjustment by health care providers on a weekly basis in the HD unit as needed. At the end of the study, both intervention and control groups will receive a home BP monitor as compensation for participation.

The baseline surveys that will be administered at initiation of the study include: 1) Modified Mini Mental State Exam (3MS) to measure global cognitive function, 2) Patient Health Questionnaire (PHQ-9) to screen and measure for depression, 3) ENRICH Social Support Instrument (ESSI) to measure the participant's level of social support, 4) BP Control in HD Knowledge Scale to measure the participant's comprehension of behaviors necessary for BP control in HD and the 5) BP Control in HD Self-efficacy Scale will be used to measure self confidence in their ability to control BP.

BP Control self-regulation measures will also be monitored and collected throughout the 12 weeks. BP control self-monitoring will be measured as adherence to recommended guidelines for monitoring in the study. To measure BP control self-evaluation and self-reinforcement, specific questions will be asked at the end of each BP and fluid log and salt check list to determine if goals were met or not met and if appropriate self-reinforcement was given.

Pre HD BPs and interdialytic weight gain (IDWG) will be collected weekly in both groups over 12 weeks. After 12 weeks the BP Control Knowledge Test, BP Control Self-Efficacy Scale, PHQ-9 and Morisky scales will be administered to both the intervention and control groups. At 30 days post intervention, the research coordinator will again collect average monthly BP and fluid gains.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years
2. average 4 week pre HD systolic BP > 150 mmHg or diastolic BP > 90 mmHg
3. read and speak English.

Exclusion Criteria:

1. on HD < 6 months
2. history of illicit drug use
3. current major depression
4. lack of orientation to person, time or place or score or < 80 on the Modified Mini Mental Status Screen
5. major health problems ie. terminal cancer or HIV
6. missed > 2 HD treatments over 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 12 weeks and 16 weeks post intervention
  Average BPs were calculated from the hemodialysis flow sheets. Pre hemodialysis BPs were averaged to determine BP at baseline, 12 weeks and 16 weeks

SECONDARY OUTCOMES:
Interdialytic Weight gain (IDWG) - Weight gain in kg between hemodialysis treatments | 12 weeks and 16 weeks post intervention
  IDWGs were calcuated by subtracting the patient's weight after their last HD treatment from weight before the next HD treatment. Three IDWGs were averaged in order to determine mean weekly IDWG

CONTACTS AND LOCATIONS:
Overall Officials: Zorica Kauric-Klein, MSN, Principal Investigator — Wayne State University
Locations (2):
- United States (2):
  - Davita Detroit Kresge Hemodialysis Unit, Detroit, Michigan
  - William Beaumont Hemodialysis Units, Royal Oak, Michigan